CLINICAL TRIAL: NCT01614782
Title: A Multiple Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK-5823 in Healthy Overweight/Obese Subjects and Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK-5823 in Overweight or Obese Participants Who Are Healthy or Have Type 2 Diabetes Mellitus (MK-5823-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5823-002
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 0.35 mg MK-5823 - Healthy Participants (Experimental)
  Interventions: Drug: MK-5823; Other: Placebo
- 0.7 mg MK-5823 - Healthy Participants (Experimental)
  Interventions: Drug: MK-5823; Other: Placebo
- 1.4 mg MK-5823 - Healthy Participants (Experimental)
  Interventions: Drug: MK-5823; Other: Placebo
- 2.8 mg MK-5823 - Healthy Participants (Experimental)
  Interventions: Drug: MK-5823; Other: Placebo
- 1.4 mg MK-5823 - Participants with T2DM (Experimental)
  Interventions: Drug: MK-5823; Other: Placebo
- 2.8 mg MK-5823 - Participants with T2DM (Experimental)
  Interventions: Drug: MK-5823; Other: Placebo

INTERVENTIONS:
Drug: MK-5823 — MK-5823 administered subcutaneously (doses ranging from 0.35 mg to 2.8 mg) once daily for 3 weeks. Doses may be adjusted downward based on safety, tolerability, and/or pharmacokinetic data. The decision to dose escalate will be based on accrued safety/tolerability data at the prior dose level.
  In each arm, 6 participants will be randomized to receive study drug and 2 participants will be randomized to receive placebo.
Other: Placebo — Matching placebo to MK-5823 administered subcutaneously once daily for 3 weeks.

SUMMARY:
The purpose of this study is to assess the multiple rising dose safety/tolerability and pharmacokinetics of MK-5823 in overweight/obese participants who are healthy and overweight/obese participants with Type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential
* A Body Mass Index between 27 and 35 kg/m^2 and weighs at least 50 kg
* Judged to be in good health and for the T2DM Panels, good health other than the diagnosis of T2DM
* For T2DM Panels only: has a diagnosis of T2DM and is being treated with lifestyle management (e.g. diet and exercise) alone or in combination with a stable dose of metformin
* A nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months

Exclusion Criteria:

* History of stroke, chronic seizures or major neurological disorder
* History of clinically significant gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
* History of clinically significant endocrine abnormalities or diseases (including type I or type II, or steroid-induced diabetes for healthy participant panel; and excluding T2DM for the T2DM Panels)
* Irritable bowel syndrome, or recurrent nausea, vomiting, diarrhea, or abdominal pain.
* History of neoplastic disease
* History of cataracts, diabetic retinopathy, macular edema, macular degeneration, vitreous hemorrhage, glaucoma, ocular surgery, ocular trauma or blindness
* Requires treatment with systemic or ocular corticosteroids
* For T2DM Panels, a history of hypoglycemic unawareness
* For T2DM Panels, active treatment with any anti-hyperglycemic drug other than metformin
* For T2DM Panels, treatment with any peroxisome proliferator-activated receptor-gamma agonist (e.g. Avandia or Actos) within 12 weeks of study participation
* Unable to refrain from using any medication beginning 2 weeks before study participation
* Consumes excessive amounts of alcohol (>3 per day)
* Consumes more than 6 caffeinated beverages per day
* Had major surgery or donated or lost more than 1 unit of blood
* Participated in another investigational study within 4 weeks of study participation
* History of significant multiple and/or severe allergies or anaphylactic reaction
* Hypersensitivity to glucagon or insulin
* Uses illicit drugs or has a history of drug or alcohol abuse within 3 months of study participation
* Woman of child-bearing potential or is a nursing mother
* For T2DM Panels, age >50 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced at least one adverse event | Up to 49 days
Number of participants who discontinued from study drug due to an adverse event | Up to 21 days

SECONDARY OUTCOMES:
Area under the plasma concentration time curve from Hour 0 to Hour 24 (AUC0-24) following once daily administration of MK-5823 | Predose on Day 1 (baseline) through 672 hours following the initial dose
Maximum plasma concentration (Cmax) following once daily administration of MK-5823 | Predose on Day 1 (baseline) through 672 hours following the initial dose
Lowest plasma concentration (Ctrough) following once daily administration of MK-5823 | Predose on Day 1 (baseline) through 672 hours following the initial dose
Time to maximum plasma concentration (Tmax) following once daily administration of MK-5823 | Predose on Day 1 (baseline) through 672 hours following the initial dose
Apparent terminal half-life (apparent t1/2) following once daily administration of MK-5823 | Predose on Day 1 (baseline) through 672 hours following the initial dose